CLINICAL TRIAL: NCT06770946
Title: The Effect of Amniotic Membrane Application on Post-Cesarean Wound Healing and Cosmetic Outcomes: a Double-Blind, Randomized Controlled Trial
Brief Title: The Effect of Amniotic Membrane Application on Post-Cesarean Wound Healing and Cosmetic Outcomes
Acronym: Amniotic Membr
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Izzet Celegen, Assistant professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/22-05
Record Dates: First submitted 2024-12-31; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Cesarean Section
Keywords: Amniotic Membrane; Cesarean Section; Wound Healing; Surgical Site Infection; Postoperative Pain; Hypertrophic Scarring; Keloid Formation; Cosmetic Outcomes; Regenerative Medicine; Maternal Health
MeSH Terms: conditions — Surgical Wound Infection; Pain, Postoperative; Cicatrix, Hypertrophic

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group design, where participants are randomly assigned to one of two groups:
  Intervention Group: Participants receive an amniotic membrane application over the cesarean incision site.
  Control Group: Participants undergo cesarean delivery without amniotic membrane application.
  Both groups were followed simultaneously to evaluate postoperative outcomes, including surgical site infection, wound healing, pain, and cosmetic satisfaction. Randomization was performed using a block randomization method to ensure balanced group sizes. This design ensures a robust comparison between the intervention and control groups under similar conditions.
Who Masked: Participant, Outcomes Assessor
Masking Description: No additional parties are masked beyond the Participant and Outcomes Assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amniotic Membrane Group (Experimental): Participants in this arm received an amniotic membrane application directly to the cesarean incision site during surgery. The membrane was harvested intraoperatively from the placenta and placed over the incision area before closure. It was removed 24 hours postoperatively, followed by standard postoperative wound care.
  Interventions: Other: Amniotic Membrane Application
- Control Group (No Intervention) (No Intervention): Participants in this arm underwent standard cesarean delivery without the application of an amniotic membrane. Standard postoperative wound care was provided without any additional intervention.

INTERVENTIONS:
Other: Amniotic Membrane Application — Amniotic Membrane Application:
  This intervention involves the application of an amniotic membrane harvested intraoperatively from the fetal side of the placenta during cesarean delivery. The membrane is placed directly on the incision site before surgical closure to promote wound healing and reduce complications such as infection, dehiscence, and scarring. The membrane is removed 24 hours postoperatively, and standard wound care is continued thereafter.
  Arms: Amniotic Membrane Group

SUMMARY:
This clinical trial evaluates the effectiveness of amniotic membrane application during cesarean delivery in reducing post-surgical complications and improving wound healing and cosmetic outcomes in women aged 18-40 undergoing their first cesarean section. The primary questions this study aims to answer are:

1. Compared to standard care, Does the amniotic membrane reduce surgical site infections and wound dehiscence?
2. Does the amniotic membrane improve patient satisfaction with cosmetic outcomes?

Participants were randomized into two groups: the intervention group received an amniotic membrane application over the cesarean incision site, while the control group underwent cesarean delivery without membrane application. Outcomes were assessed at predefined postoperative intervals, focusing on wound healing, pain levels, and cosmetic satisfaction.

DETAILED DESCRIPTION:
This randomized, double-blind, controlled trial investigates the effectiveness of amniotic membrane application in reducing post-cesarean complications, including surgical site infections, wound dehiscence, and scar formation. The trial also assesses its impact on pain management and cosmetic outcomes in women aged 18-40 undergoing their first cesarean section. The study was conducted between May 2022 and May 2023 at Van Regional Training and Research Hospital.

The amniotic membrane, the innermost layer of the placenta, has regenerative, anti-inflammatory, and antimicrobial properties. Its application during cesarean delivery may offer a cost-effective and autologous intervention to enhance surgical outcomes and patient satisfaction.

Objectives:

Primary Objectives:

1. Evaluate whether the amniotic membrane reduces surgical complications, including infections, hematoma, and wound dehiscence.
2. Investigate its role in preventing hypertrophic scars and keloids.

Secondary Objectives:

1. Assess the effect of amniotic membrane application on postoperative pain levels using the Visual Analog Scale (VAS).
2. Measure patient satisfaction with cosmetic results using the Modified Hollander Wound Evaluation Scale.

Methodology:

A total of 372 participants were enrolled and randomized into two groups (1:1 ratio) using block randomization to ensure balanced allocation. The intervention group received an amniotic membrane, harvested intraoperatively from the placenta and applied directly to the cesarean incision site before closure. The control group underwent cesarean delivery without membrane application. Both groups were blinded to their assignments, and standard postoperative wound care was provided.

Participants were evaluated at multiple predefined postoperative time points (days 1, 2, 7, 40, and 6 months) for surgical site infections, wound dehiscence, scar/keloid formation, pain levels, and cosmetic satisfaction.

Significance:

This study provides evidence supporting the use of autologous amniotic membranes in obstetrics, potentially establishing a low-cost, accessible method to improve surgical outcomes and patient quality of life. If successful, these findings may have broader implications for other surgical fields and high-risk patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18-40 years. Undergoing their first cesarean section. Term pregnancies (≥37 weeks of gestation). Elective cesarean delivery performed under spinal anesthesia. Use of the Pfannenstiel incision method. Willing and able to provide written informed consent.

Exclusion Criteria:

* History of previous abdominal surgeries. Presence of chronic conditions such as diabetes mellitus, hypertension, or vascular diseases.

Pulmonary conditions or collagen tissue disorders affecting wound healing. Signs of infection during delivery. Use of medications or therapies that impair wound healing (e.g., corticosteroids, immunosuppressants).

Known hypersensitivity to materials or methods used in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study is limited to individuals with a biological sex of female, as it involves cesarean delivery outcomes
Enrollment: 372 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection (SSI) | Time Frame: Within 7 days post-surgery.
  Description: The presence of surgical site infections diagnosed based on erythema, induration, tenderness, and purulent discharge.
  Scale: Binary (Yes/No)
Wound Dehiscence | Time Frame: Within 7 days post-surgery.
  Description: The occurrence of wound dehiscence defined as a wound gap of less than 1 cm in depth.
  Scale: Binary (Yes/No).
Scar/Keloid Formation | Time Frame: At 40 days and 6 months post-surgery.
  Description: The presence of hypertrophic scars or keloids assessed visually. Scale: Binary (Yes/No).

SECONDARY OUTCOMES:
Postoperative Pain (VAS Score) | Time Frame: Postoperative days 1 and 2.
  Description: Pain scores measured using the Visual Analog Scale (VAS). Scale: 0 to 10 (0 = no pain, 10 = worst pain).
Cosmetic Satisfaction | Time Frame: At 40 days post-surgery.
  Description: Patient-reported satisfaction with the cosmetic appearance of the incision site, measured using the Modified Hollander Wound Evaluation Scale.
  Scale: 0 to 6 (higher scores indicate better cosmetic outcomes).

CONTACTS AND LOCATIONS:
Locations (1):
- Van Regional Training and Research Hospital, Van, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Plan to Share IPD: No Plan Description: Individual participant data will not be shared due to institutional data-sharing policies and privacy concerns.